CLINICAL TRIAL: NCT05612048
Title: Pilot Study of Dental Erosion as a Non-invasive Biomarker of Esophagogastric Cancer
Brief Title: A Study of Tooth Erosion in People With Esophagogastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-370
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Esophagogastric Cancer
Keywords: Tooth erosion; GERD; Loss of tooth enamel; 22-370
MeSH Terms: conditions — Tooth Erosion; Gastroesophageal Reflux | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Patients will complete a questionnaire and undergo imaging by the intra-oral camera of their teeth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients diagnosed with esophagogastric cancer (Experimental): Patients have completed the intervention once completing the survey, undergoing dental imaging and future patients will also provide an optional saliva sample.
  Interventions: Other: Survey; Other: Intra-oral camera; Other: Optional Salvia sample
- Patients diagnosed with colorectal, pancreatic, breast, head and neck, or non-small cell lung cancer (Experimental): Patients undergo consenting and dental imaging during their routine visits at MSK.
  Interventions: Other: Survey; Other: Intra-oral camera
- Healthy volunteers who have not been diagnosed with cancer (Experimental): Healthy controls will be defined as those without a known or suspected invasive cancer history and excluding those undergoing a procedure for symptomatic reflux.
  Interventions: Other: Survey; Other: Intra-oral camera

INTERVENTIONS:
Other: Survey — This is a 15-item questionnaire. The questionnaire asks subjects to quantify, during a specified duration of time, the number of times they have consumed or completed a task (ex. alcohol intake, cigarette use, and teeth brushing frequency). Additionally, the questionnaire further asks subjects to quantify their GERD symptoms and risk factors prior to diagnosis. All study procedures will be completed in one visit as part of a standard-of-care clinic visit.
Other: Intra-oral camera — Intraoral pictures of molars and incisors in 13 key regions
Other: Optional Salvia sample — Cohort 1 only. Participant is responsible for collecting and bringing the salvia sample to clinic.
  Arms: Patients diagnosed with esophagogastric cancer

SUMMARY:
The researchers are doing this study to find out more about what may lead to the loss of tooth enamel (the thin outer covering of the tooth) and how often it happens in people with esophagogastric cancer, colorectal cancer, pancreatic cancer, breast cancer, head and neck cancer, or non-small cell lung cancer, or a healthy volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to provide written informed consent.
* Patients with a history of esophagogastric, HNSCC, PDAC, CRC, or NSCLC or healthy controls
* Patients must be able to fully comprehend and complete the survey and be willing to have pictures taken of their teeth with a camera or intra-oral camera.
* Patients must be able to understand English language or have access to adequate translation services.
* Age ≥ 18 years old.

Exclusion Criteria:

* Subjects without evaluable molars or with significant molar dental work precluding dentists from assessing enamel status, Note: evaluable is defined as having bilateral assessable mandibular molars, or erosions present in the remaining assessable quadrants.
* For healthy controls only, patients cannot have a non-skin cancer history nor presenting for a procedure evaluating reflux symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The incidence of dental erosions | 1 year
  scored with a modified BEWE index.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Maron, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm